CLINICAL TRIAL: NCT06320145
Title: Effect of Cryotherapy on Primary Dysmenorrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marslino Mohsen Beshrida, Resident of Physical Therapy for Woman's Health Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004045
Record Dates: First submitted 2023-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Dysmenorrhea Primary
Keywords: Cryotherapy; Primary dysmenorrhoea
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Cryotherapy Group) (Experimental): About 15 Women suffering from primary dysmenorrhoea who will receive cryotherapy sessions (3 days per week for 20 minutes), in addition to core stability exercise.
  Interventions: Device: Cryotherapy; Other: core stability exercises
- Group B (core stability Group) (Experimental): About 15 Women suffering from primary dysmenorrhoea who will receive core stability exercises only
  Interventions: Other: core stability exercises

INTERVENTIONS:
Device: Cryotherapy — This device used at the first, second and third day of period to decrease pain for 20 min at first, second and third day
  Arms: Group A (Cryotherapy Group)
Other: core stability exercises — core stability exercises

SUMMARY:
Dysmenorrhea is a menstrual disorder defined by the presence of painful cramps of uterine origin that occur during menstruation. It is one of the most common causes of pelvic pain and short-term absenteeism from school or work, among young and adult women.

Cryotherapy, therapeutic cooling, is one of the modalities widely used in sports medicine for a variety of treatment purposes. Physiological and neurological responses of musculoskeletal tissues to cooling have been extensively examined in the literature.

DETAILED DESCRIPTION:
Dysmenorrhea is an existing mainstream gynecologic problem which habitually affects females of reproductive age.

Dysmenorrhea is of two types: Primary dysmenorrhea and secondary dysmenorrhea :.

primary dysmenorrhea is painful menstrual cramps without any evident pathology to account for them, and it occurs in up to 50% of menstruating females and causes significant disruption in quality of life and absenteeism.

The main cause of primary dysmenorrhea is prostaglandin production. This is naturally present substance that is made by uterine cells. It helps in contraction of the muscles, thus assisting in shedding of the uterine lining every month. When the production of prostaglandin is high, it leads to excessive pain and cramps. The prostaglandin is the main cause of other symptoms associated with primary dysmenorrhea, like nausea and vomiting.

Dysmenorrhea has a negative effect on a woman's life. It may be so severe as to confine the woman to bed during adolescence, dysmenorrhea leads to high rates of absence from school and non-participation in activities. Mild to moderate cases can usually be treated by reassurance and paracetamol

Cryotherapy, a physical therapy modality, is widespread in clinical rehabilitation practice for the management of the inflammatory phase of tissue repair. It can decrease tissue temperature and subsequently reduce inflammatory symptoms such as pain and swelling. Generally, the mechanisms underlying the reduction of inflammatory symptoms by cryotherapy are associated with a decrease in tissue temperature and reduction of vasopermiability, blood flow, nerve conduction velocity, and cell metabolism .

Core stability exercise has been known as a beneficial intervention in the management of several medical prob- lems. Core stability exercises strengthen and coordinate the muscles around the abdominal, lumbar, and pelvic regions Because it has been suggested that the core stability exercises mainly affect the lumbosacral muscles and increase blood supply in lumbosacral structures .

the purpose of core strengthening is to combine the concepts of lumber stabilization and how instability can lead to injury and pain specifically during stressful times of the female body and one of these repetitive stressful times is dysmenorrhea.

The lumber portion of spine is sturdy and designed to take the force of the body and it also involved in the origin and insertion of certain musculature and nerve innervations to their correlated areas. If at any time a certain part of the lumbar spine is weak, it is not as its optimal level to handle functional stress, which can result in pain throughout the abdomen, low back, or thighs. These areas just happen to be the same areas that are affected by females suffering from dysmenorrhea

Core strengthening allows the small intrinsic musculature surrounding the lumbar spine to be conditioned for greater performance, this type of training allows for isolation and strengthening of core muscle groups. When these muscles are strong, they are much more prepared to handle daily forces of normal biomechanics, even when the body is under the stress of the menstrual cycle , Core strengthening is a description of the muscular control around the lumbar spine to maintain functional stability.

ELIGIBILITY:
Inclusion Criteria:

* All females with moderate to severe primary dysmenorrhea (as determined by V.A.S and WaLIDD Scale).
* All females will be virginal and non-smokers.
* Their BMI will be range from 20-30 kg/m2.
* They have regular menstrual cycle with menstrual cycle length of 28-30 days.

Exclusion Criteria: (patients will be excluded if they had):

* Any Pelvic pathology
* Malignancy.
* Uncontrolled type l Diabetes.
* Epilepsy
* pacemaker
* cancer
* skin disease

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Pain assessed by VAS | 2 months
  Pain which is assessed by VAS scale ( which is from 0 to 10 the VAS as being 10 cm horizontal line with one end described as (no pain =0), and other end (the worst pain I ever felt = 10). Patients will be asked to mark a point on the line between the extremes that relates to their level of pain

CONTACTS AND LOCATIONS:
Overall Officials: SOHAIR ELKOSAIRY, Professor, Study Chair — Chairman of Physical Therapy,Faculty of Physical Therapy,Cairo University
Locations (1):
- Faculty of Physical Therapy,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No